CLINICAL TRIAL: NCT01479803
Title: COMPARATIVE STUDY OF DIAGNOSTIC VALUE FOR THE ECHOTIP® PROCORE™ 22 Gauge NEEDLE VERSUS ECHOTIP® 22 Gauge IN THE DIAGNOSIS OF PANCREATIC SOLID TUMORS UNDER ENDOSCOPIC ULTRASONOGRAPHY : THE "PICORE" STUDY
Brief Title: Comparison of Two Needles (ProCore vs EchoTip) for the Diagnosis of Pancreatic Solid Mass Under EUS
Acronym: PICORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VANBIERVLIET (Other)
Responsible Party: Sponsor-Investigator, VANBIERVLIET, Director, Head of endoscopy, Principal Investigator, Medical doctor, Société Française d'Endoscopie Digestive
Organization: Société Française d'Endoscopie Digestive (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2011-A00578-33
Record Dates: First submitted 2011-10-20; First posted 2011-11-24 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Pancreatic Tumor; Fine Needle Aspiration; Endoscopic Ultrasonography
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Punctures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EchoTip HD ProCore 22 Gauge (Active Comparator): first passage in the pancreatic tumor with the EchoTip HD ProCore 22 Gauge then with the EchoTip 22 Gauge
  Interventions: Procedure: Puncture with fine needle aspiration under endoscopic ultrasonographic control
- Echo Tip 22 Gauge (Active Comparator): First passage through the tumor with the EchoTip 22 Gauge then with Echotip HD ProCore 22 Gauge
  Interventions: Procedure: Puncture with fine needle aspiration under endoscopic ultrasonographic control

INTERVENTIONS:
Procedure: Puncture with fine needle aspiration under endoscopic ultrasonographic control — Puncture of the pancreatic solid mass with fine needle aspiration under endoscopic ultrasonographic control Passage in the same pancreatic mass of first EchoTip HD Procore then EchoTip 22 Gauge or vice versa according to the randomization

SUMMARY:
The negative predictive value of fine needle aspiration under ultrasound endoscopy (EUS) for the diagnostic of solid pancreatic masses is 70% on average in the current literature with 22 gauge needles. There is a wide variability of this rate across studies (from 38 to 92%). In case of negativity of the biopsy, the risk of missing a pancreatic cancer whose prognosis is severe and extensive treatment, remains important. To improve the sensitivity of EUS echo endoscopy, several methods were used. A new needle (Echo Tip ® HD ProCore ™) has received CE Mark in the field of EUS. This instrument combines the comfortable and handy size of 22 Gauge and innovative design (window lateralized bevel) with in vitro studies obtaining core biopsy. In addition, a single pass through the tumor is achieved with this hand against several (2-3 minimum) with the current hardware. The theoretical goal is to have a tissue material more abundant during the sampling, without increasing morbidity and increase the diagnostic accuracy. A preliminary prospective study with this material has shown interesting results (increase the diagnostic accuracy of 15%).

To determine the diagnostic gain with this new hand, it seemed essential to propose a prospective comparative study (22 gauge needle ProCore ™ versus the old EchoTip ® 22-Gauge) randomized (randomization of the order of the needles) in crossover (on the same lesion) in samples of pancreatic solid tumors. The caliber of 22 gauge is the gauge most often used for punctures under ultrasound endoscopy, resulting in less morbidity. Puncture by the 2 needles on the same injury can limit the effect of variability between patients and thereby have a better power for the investigators study without increasing the risk of complications (the needle ProCore ™ does not require that one pass through the tumor). The study of pancreatic solid tumors is one that poses the biggest diagnostic problem still present in the investigators daily practice. The aim of this study is to compare the diagnostic accuracy of the needle ProCore™ versus EchoTip® in etiological cyto histological diagnostic for pancreatic solid tumors under EUS.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor of the pancreas (<50% share or anechoic fluid) to receive a biopsy under endoscopic ultrasonography (EUS)

Exclusion Criteria:

* Contraindications to the achievement of an upper gastrointestinal endoscopy
* Haemorrhagic disease, disorder of hemostasis and coagulation (PT <60%, CaT> 40 sec. and platelets <60000/mm3)
* Pancreatic cystic mass (fluid quota valued at more than 50% of the mass lesion on imaging)
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of fine needle aspiration Echo Tip® HD ProCore™ versus EchoTip® in the etiological cyto histological in pancreatic solid tumors explored under endoscopy ultrasonography. | 6 months

SECONDARY OUTCOMES:
Immediate morbidity per procedure of both techniques and delayed morbidity (up to D30) of the complete procedure (corresponding to all of the discussion with the punctures of 2 needles). | 2 minutes and 30 days
  Adverse effects (%, number of event for each needle passage) during the procedure or during the follow up period (30 days)
Quality of histological specimen obtained with the 2 needles | 10 days
  Visual analogic scale and Maier score used for this point
Dysfunction in two type of needle biopsy | Day one
  failure or difficulty reports with each needle (%)
ease of puncture between the 2 types of equipment. | day one
  Visual analogic scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital L'Archet 2, CHU Nice, BP 3079, Nice, France

REFERENCES:
- [Derived] Vanbiervliet G, Napoleon B, Saint Paul MC, Sakarovitch C, Wangermez M, Bichard P, Subtil C, Koch S, Grandval P, Gincul R, Karsenti D, Heyries L, Duchmann JC, Bourgaux JF, Levy M, Calament G, Fumex F, Pujol B, Lefort C, Poincloux L, Pagenault M, Bonin EA, Fabre M, Barthet M. Core needle versus standard needle for endoscopic ultrasound-guided biopsy of solid pancreatic masses: a randomized crossover study. Endoscopy. 2014 Dec;46(12):1063-70. doi: 10.1055/s-0034-1377559. Epub 2014 Aug 6. PMID 25098612